CLINICAL TRIAL: NCT06249191
Title: A Phase Ib/II Study Evaluating the Safety and Efficacy of Mosunetuzumab in Combination With DA EPOCH in Previously Untreated C-Myc Rearrangement Positive High-Grade B Cell Lymphomas
Brief Title: Mosunetuzumab With Chemotherapy for the Treatment of Patients With Untreated C-Myc Rearrangement Positive High Grade B Cell Lymphoma or Diffuse Large B Cell Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Genentech, Inc. (Industry); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Stephen Spurgeon, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00023707; NCI-2024-00070 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00023707 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Diffuse Large B-Cell Lymphoma; High Grade B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Biopsy; Specimen Handling; Cyclophosphamide; Doxorubicin; Etoposide; Magnetic Resonance Spectroscopy; Prednisone; deltacortene; prednylidene; Vincristine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Mosunetuzumab and EPOCH) (Experimental): Patients receive mosunetuzumab IV, over 2-4 hours, on day 1, 8 and 15 of cycle 1 and day 1 of subsequent cycles. Patients receive etoposide IV, doxorubicin IV, and vincristine IV on days 1-4, cyclophosphamide IV, over 2 hours, on day 5 and prednisone PO BID on days 1-5 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity for up to 6 cycles. Patients undergo bone marrow aspiration and biopsy, tumor biopsy and may undergo echocardiography or MUGA at screening and PET scan, CT scan or MRI and blood sample collection throughout the study.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration and Biopsy; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Doxorubicin; Procedure: Echocardiography; Drug: Etoposide; Procedure: Magnetic Resonance Imaging; Biological: Mosunetuzumab; Procedure: Multigated Acquisition Scan; Procedure: Positron Emission Tomography; Drug: Prednisone; Drug: Vincristine

INTERVENTIONS:
Procedure: Biopsy — Undergo tumor biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration and Biopsy — Undergo bone marrow aspiration and biopsy
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B-518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719; WR-138719
Drug: Doxorubicin — Given IV
  Other Names: Adriablastin; Hydroxydaunomycin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
Procedure: Echocardiography — Undergo echocardiography
  Other Names: EC
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP 16213; VP-16; VP-16-213; VP16
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Mosunetuzumab — Given IV
  Other Names: Anti-CD20 x Anti-CD3 Bispecific Monoclonal Antibody BTCT4465A; BTCT 4465A; BTCT-4465A; BTCT4465A; CD20/CD3 BiMAb BTCT4465A; Lunsumio; Mosunetuzumab-axgb; RG 7828; RG-7828; RG7828; RO7030816
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Drug: Vincristine — Given IV
  Other Names: LCR; Leurocristine; VCR; Vincrystine

SUMMARY:
This phase Ib/II clinical trial tests the safety, side effects, and effectiveness of mosunetuzumab with chemotherapy for the treatment of patients with untreated, c-Myc rearrangement positive, high grade B cell lymphoma or diffuse large B cell lymphoma. A monoclonal antibody is a type of protein that can bind to certain targets in the body, such as molecules that cause the body to make an immune response (antigens). Immunotherapy with monoclonal antibodies, such as mosunetuzumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Chemotherapy drugs, such as etoposide, doxorubicin, vincristine, cyclophosphamide and prednisone work in different ways to stop the growth of cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving mosunetuzumab with chemotherapy may be safe, tolerable and/or effective in treating patients with untreated, c-Myc rearrangement positive, high grade B cell lymphoma or diffuse large B cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the safety and tolerability of the mosunetuzumab (M) plus dose-adjusted (DA) etoposide, doxorubicin, vincristine, cyclophosphamide, and prednisone [EPOCH] combination in previously untreated c-Myc + high-grade B cell lymphoma. (Phase Ib) II. Evaluate the efficacy of M DA EPOCH as complete response (CR) in previously untreated c-Myc + high grade B cell lymphoma. (Phase II)

SECONDARY OBJECTIVES:

I. Evaluate the efficacy of M DA EPOCH in Phase Ib and II as overall response, durability of response, and survival.

II. Ongoing evaluation of the toxicity and tolerability of M DA EPOCH. (Phase Ib and II) III. Summarize DA EPOCH treatment details when received as part of M DA EPOCH. (Phase Ib and II)

EXPLORATORY OBJECTIVES:

I. Assess utilization and benefit of tocilizumab for toxicity management. (Phase Ib and II) II. Assess toxicity of M DA EPOCH based on immune related AEs (irAEs). (Phase Ib and II) III. Identify baseline factors of response and progression. (Phase Ib and II) IV. Assess the immune response to mosunetuzumab in the setting of the M DA EPOCH regimen. (Phase Ib and II)

OUTLINE:

Patients receive mosunetuzumab intravenously (IV), over 2-4 hours, on day 1, 8 and 15 of cycle 1 and day 1 of subsequent cycles. Patients receive etoposide IV, doxorubicin IV, and vincristine IV on days 1-4, cyclophosphamide IV, over 2 hours, on day 5 and prednisone orally (PO) twice per day (BID) on days 1-5 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity for up to 6 cycles. Patients undergo bone marrow aspiration and biopsy, tumor biopsy and may undergo echocardiography or multigated acquisition scan (MUGA) at screening and positron emission tomography (PET) scan, computed tomography (CT) scan or magnetic resonance imaging (MRI) and blood sample collection throughout the study.

After completion of study treatment, patients are followed up every 3 months for 2 years then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* For both phases of the study, participant must be 18-75 years of age and have previously untreated high-grade B cell lymphoma (HGBCL) or diffuse large B cell lymphoma (DLBCL), including transformed DLBCL per the World Health Organization (WHO) 2022 classification, and with documented c-Myc rearrangement on fluorescence in situ hybridization (FISH) testing. Eligible types of c-Myc rearrangements will be performed by FISH testing and may include any single MYC rearrangement (single-hit lymphoma), Double hit (DHL) lymphoma or and triple hit (THL) lymphoma defined by translocations of MYC and BCL2 (DHL) and BCL6 (THL)
* Pathology must be verified and confirmed by university pathologists at the enrolling institution and centrally (OHSU) for any biopsies read outside of either institution
* Stage II or higher and International Prognostic Index (IPI) score of 2-5
* Able to comply with the study protocol and procedures, in the investigator's judgment
* At least one bi-dimensionally measurable nodal lesion, defined as ≥ 1.5 cm in its longest dimension, or one bi-dimensionally measurable extranodal lesion, defined as ≥ 1.0 cm in its longest diameter
* Confirmed availability of archival or freshly collected tumor tissue before study enrollment
* Eastern Cooperative Oncology Group Performance Status of 0, 1, or 2
* Left ventricular ejection fraction (LVEF) defined by multiple-gated acquisition (MUGA) scan or echocardiogram (ECHO) within the institutional limits of normal
* Absolute neutrophil count (ANC) ≥ 1.0 ×10^9/L (14 days prior to first mosunetuzumab dose) (unless inadequate function is due to underlying disease, as established by extensive bone marrow involvement, or is due to hypersplenism secondary to the involvement of the spleen by lymphoma per the investigator) without transfusion
* Platelet count ≥ 75 ×10^9/L (14 days prior to first mosunetuzumab dose) (unless inadequate function is due to underlying disease, as established by extensive bone marrow involvement, or is due to hypersplenism secondary to the involvement of the spleen by lymphoma per the investigator) without transfusion
* Total hemoglobin ≥ 10 g/dL (21 days prior to first mosunetuzumab dose) (unless inadequate function is due to underlying disease, as established by extensive bone marrow involvement, or is due to hypersplenism secondary to the involvement of the spleen by lymphoma per the investigator) without transfusion
* Serum creatinine ≤ upper limit of normal (ULN); or estimated creatinine clearance ≥ 50 mL/min by Cockcroft Gault method or other institutional standard methods, e.g. based on nuclear medicine renal scan
* For persons of childbearing potential (PCBP), an agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of < 1% per year, and confirmed agreement to refrain from donating eggs, during the treatment period and for at least 3 months after the last dose of mosunetuzumab, and 3 months after the last dose of tocilizumab (if applicable), whichever is longer
* For participants who can produce sperm and create pregnancy: confirmed agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm

Exclusion Criteria:

* Pregnant or breast /chestfeeding
* Prior treatment for DLBCL. Exceptions:

  * Prednisone of ≤ 100 mg for up to 10 days, within 28 days prior to starting study treatment. Prednisone or equivalent corticosteroid must be discontinued by the time of treatment start
  * One cycle of RCHOP or DA R EPOCH
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies or known sensitivity or allergy to murine products
* Contraindication to receive full dose of any of the individual components of EPOCH
* Participants with history of confirmed progressive multifocal leukoencephalopathy (PML)
* Known or suspected chronic active Epstein Barr virus (CAEBV) infection
* Positive test results for chronic hepatitis B infection (defined as positive hepatitis B surface antigen [HBsAg] serology)

  * Participants with occult or prior hepatitis B infection (defined as positive total hepatitis B core antibody and negative HBsAg) may be included if hepatitis B virus (HBV) deoxyribonucleic acid (DNA) is undetectable at the time of screening. These Participants must be willing to undergo monthly DNA testing and appropriate antiviral therapy as indicated
* Acute or chronic hepatitis C virus (HCV) infection. Participants positive for HCV by antibody testing, but negative for HCV by polymerase chain reaction (PCR) are eligible
* HIV seropositivity
* Administration of a live, attenuated vaccine within 4 weeks before first study treatment administration or anticipation that such a live, attenuated vaccine will be required during the study
* Prior solid organ transplantation
* Known or suspected history of hemophagocytic lymphohistiocytosis (HLH).
* History of autoimmune disease, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis. Exceptions:

  * Participants with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone may be eligible.
  * Participants with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
  * Participants with a history of disease-related immune thrombocytopenic purpura, autoimmune hemolytic anemia, or other stable autoimmune diseases may be eligible after review and approval by the primary investigator (PI)
* Systemic immunosuppressive medications (including, but not limited to, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents) with the exception of pre-phase treatment with prednisone up to 100 mg daily for 7 days (or equivalent corticosteroid dose) prior to cycle 1 day 1 (C1D1). Exceptions:

  * The use of inhaled corticosteroids is permitted.
  * The use of mineralocorticoids for management of orthostatic hypotension is permitted.
  * The use of physiologic doses of corticosteroids for management of adrenal insufficiency is permitted
* Current active central nervous system (CNS) involvement of lymphoma on the screening MRI brain
* Current or past history of CNS disease, such as stroke, epilepsy, CNS vasculitis, neurodegenerative disease. Exceptions:

  * Participants with a history of stroke who have not experienced a stroke or transient ischemic attack in the past 2 years and have no residual neurologic deficits as judged by the investigator are allowed.
  * Participants with a history of epilepsy who have had no seizures in the past 2 years while not receiving any anti-epileptic medications are allowed in the expansion cohorts only
* Prior radiotherapy to the mediastinal / pericardial region within 4 weeks
* Malignancy treated with curative intent unless in documented remission without treatment for 2 years prior to enrollment, or other malignancy that could affect compliance with the protocol or interpretation of results. Exception: Participants with a history of curatively treated basal or squamous cell carcinoma or melanoma of the skin or in situ carcinoma of the cervix are eligible. Adjuvant endocrine therapy for non-metastatic, hormone receptor-positive breast cancer is permitted
* Evidence of significant, uncontrolled concomitant diseases that could affect compliance with the protocol or interpretation of results or that could increase risk to the Participant, including renal disease that would preclude chemotherapy administration or pulmonary disease (including obstructive pulmonary disease and history of bronchospasm)
* Significant pulmonary disease (including obstructive pulmonary disease and history of bronchospasm)
* Significant cardiovascular disease, defined as

  * New York Heart Association [NYHA] Class III or IV cardiac disease,
  * Congestive heart failure,
  * Myocardial infarction within the previous 6 months,
  * Unstable arrhythmias, or
  * Unstable angina
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment or any major episode of infection requiring treatment with IV antibiotics or hospitalization (relating to the completion of the course of antibiotics) within 4 weeks before C1D1
* Clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis
* Aspartate aminotransferase (AST) or Alanine aminotransferase (ALT) > 2.5 x ULN within 14 days of initiation of study treatment
* Total bilirubin ≥ 1.5 x ULN within 14 days of initiation of study treatment
* International normalization ratio (INR) > 1.5 x ULN in the absence of therapeutic anticoagulation within 14 days of initiation of study treatment
* Partial prothrombin time (PTT) or adjusted partial prothrombin time (aPTT) > 1.5 x ULN in the absence of a lupus anticoagulant within 14 days of initiation of study treatment
* Herbal therapies intended as treatment of lymphoma
* Medicinal or recreational cannabis products are not permitted while receiving the study intervention.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-13 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) (phase Ib) | From the first dose of mosunetuzumab to the end of cycle 2 (1 cycle = 21 days)
  Using a modified 3+3 design in previously untreated c-Myc rearranged aggressive B cell lymphomas during the safety run-in period (cycle 1-2). Incidence of DLTs will be tabulated by dose level. All DLTs will be coded by system organ class, MedDRA preferred term, and severity grade using Common Terminology Criteria for Adverse Events (CTCAE )(version [v] 5.0). Cytokine Release Syndrome/Immune Effector Cell-Associated Neurotoxicity Syndrome (CRS/ICANS) toxicities will be graded with the American Society for Transplantation and Cellular Therapy (ASTCT) system. Safe dose of mosunetuzumab (or dose adjusted [DA] etoposide, doxorubicin, vincristine, cyclophosphamide, and prednisone [EOPCH]) will be specified.
Proportion of patients with complete response by positron emission tomography-computed tomography (PET-CT) (phase II) | Up to 5 years
  Will be reported with exact 95% confidence interval.

SECONDARY OUTCOMES:
Overall response rate (ORR) by PET-CT | Up to 5 years
  ORR defined as the proportion of participants who achieve a complete response (CR) or partial response (PR) among all efficacy evaluable participants by the EOT disease assessment. Will be reported with exact 95% confidence interval, by mosunetuzumab dose level if applicable.
Duration of response (DOR) | From first documented evidence of documented CR or PR to first occurrence of disease progression as determined by the investigator, or death from any cause, whichever occurs first, assessed up to 5 years
  Descriptive statistics such as median DOR, with minimum and maximum DOR, will be reported by mosunetuzumab dose level if applicable.
Progression free survival (PFS) | From the first dose of mosunetuzumab to first occurrence of disease progression or relapse as determined by the investigator, or death from any cause, whichever occurs first, assessed up to 5 years
  Are estimated in the efficacy set using the Kaplan Meier method. We will report median PFS and corresponding 95% confidence interval for participants by mosunetuzumab dose level if applicable.
Overall survival (OS) | From first dose of mosunetuzumab to death by any cause, assessed up to 5 years
  Are estimated in the efficacy set using the Kaplan Meier method. We will report median OS and corresponding 95% confidence interval for participants by mosunetuzumab dose level if applicable.
Incidence of ≥ grade 3 toxicities possibly or definitely related to mosunetuzumab | Up to to 30 days after last dose of mosunetuzumab
  Per ASTCT for CRS and ICANS;CTCAE v5.0 otherwise
Number of cycles completed and dose received of DA EPOCH | Up to to 30 days after last dose of DA EPOCH

CONTACTS AND LOCATIONS:
Overall Officials: Stephen E Spurgeon, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States